A clinical prospective study to validate a risk scoring model for the hepatic metastases from gastric cancer after curative surgery (DJY003 Trail)

**Edition Number: 1.0** 

**Edition Generation Date:** Apr 29, 2023

Principal Investigator: Jingyu Deng

Research Institute: Cancer Hospital & Institute of Tianjin Medical University

ClinicalTrials.gov ID: NCT06023966

## **Statistical Analysis Plan**

Continuous variables will be presented as mean  $\pm$  standard deviation or median (interquartile range). Statistical analyses will be performed using the Chi-square test or Fisher's exact test for the categorical variables and the T test or Mann–Whitney U test for the continuous variables. The sensitivity, specificity, PPV and NPV of the model, and the consistency between actual results of postoperative hepatic metastases occurrence and predicted results from the model will be calculated. In addition, the AUROC will be calculated to validate the calibration ability of the risk scoring model. A *p*-value threshold of 0.05 will be considered statistically significant. All statistical analyses will be performed using SPSS 26.0 software and R software.